CLINICAL TRIAL: NCT01132339
Title: Prospective Clinical Trial to Investigate Adverse Reactions to MR and CT-examinations (Enhanced and Unenhanced)
Brief Title: Adverse Reactions to MR and CT-examinations (Enhanced and Unenhanced)
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: H-1-2010-011
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Renal Adverse Events - Contrast Induced Nephropathy (CIN); Non-renal Adverse Events
Keywords: Adverse reactions to Gadolinium-based contrast agents.; Adverse reactions to Iodine-basedcontrast agents.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Enhanced MR (case group): those with an exposure to gadolinium-based contrast agent
- Unenhanced MR (control group): those without an exposure to gadolinium-based contrast agent
- Unenhanced CT (control group): those without an exposure to iodine-containing contrast agent
- Enhanced CT (case group): those with an exposure to iodine-containing contrast agent

SUMMARY:
Rationale:

Contrast agents are important tools for MR/CT- examinations, when it comes to diagnosing diseases. But despite their frequent use in Denmark, they are not free of serious and potentially fatal adverse reactions. Examples of this are contrast-induced nephropathy (CIN) and nephrogenic systemic fibrosis (NSF). Therefore, it is extremely important to clarify if these adverse reactions are actually directly related to the use of contrast agents or to MR/CT- examinations.

Objective:

To prospectively assess the incidence of adverse reactions of iodine-containing CT and gadolinium- based MR contrast agents in a prospective design. A control group examined without the use of contrast agent will be included, so that the study can illuminate reported adverse events related to contrast agents and CT/MR- examinations. This project will in the long term mean that, any significant and life-threatening delayed adverse reactions will be discovered earlier and hence it will be more likely to treat the patients in good time for these adverse reactions.

The following series of hypotheses will be investigated in this study:

1. Renal as well as non-renal adverse reactions occurring are related to the use of contrast agent in MR-/CT-examination.
2. CIN occurs in patients undergoing a MR-/CT-examination with contrast agent.

Methods:

Approvals are obtained from The Copenhagen County Committee on Biomedical Research Ethics and Danish Data Protection Agency. A total of 1600 patients will be included from Department of Radiology at Herlev Hospital, where all the MR- and CT examinations will be performed. Patients will be divided into four groups (a, b, c and d) with 400 patients in each group. Group a and c (case group) undergo respectively MR and CT examination with contrast agent While group b and d (control group) will undergo respectively MR and CT examination without the use of contrast agent. For each patient the following will be recorded: Risk factors, renal function (eGFR) before and 72 hours after MR/CT- examination as well as the incidence of immediate reactions (within 30 min.). Furthermore, patients have to answer a questionnaire 72 hours and 1 month after MR/CT- examination about the severity and frequency of adverse reactions to contrast media.

DETAILED DESCRIPTION:
Rationale and objectives:

Contrast agents continue to cause concern among patients and doctors because of their widespread use and the rare but potentially important adverse reactions associated with them. Intravenous (into a vein) contrast agents are used daily for both Computed Tomography (CT) and Magnetic Resonance (MR) examinations as an aid for detection and characterization of diseases. Despite their use for millions of examinations each year, the contrast agents are not entirely free of serious and potentially life-threatening adverse reactions. Therefore, the application of both iodine-containing and gadolinium-based contrast agents, respectively for CT and MR- examinations has raised some safety concerns, especially in patients in certain risk groups, e.g. patients with previous allergic reactions to gadolinium and iodine-containing contrast agents, patients with pre-existing renal impairment and diabetes patients. Adverse reactions of contrast agents can be divided into non-renal and renal adverse reactions. The non-renal adverse reactions may be acute or delayed. The acute adverse reactions occur within one hour after the contrast agent is administered to the patient, while the delayed adverse reactions occur after one hour and within a week.Some reactions such as Nephrogenic Systemic Fibrosis (NSF) may occur even later and is classified as a very late adverse reaction. Patients at high risk group should be identified before contrast agent administration to avoid these adverse reactions. Adverse reactions using iodine-containing contrast agents have been known for over 20 years. They are mostly mild or moderate skin reactions that occur during the period 1 hour to 7 days after contrast agent administration, and usually disappear within 3-7 days. Nevertheless, serious and life-threatening adverse reactions occur, and one of the most serious effects is Contrast Induced Nephropathy (CIN), which is a renal adverse reaction. CIN refers to a reduction in the renal function induced by contrast agent. This implies a deterioration in renal function (an increase in serum creatinine by more than 25% or 44μmol / L) occurring within three days after intravascular administration of iodine-containing contrast agent. CIN is a well known complication when it comes to radiological studies using iodine-containing contrast agents. The rapid development and frequent use of CT- examination with simultaneous administration of relatively large doses of iodine-containing contrast agents have contributed to a growing number of cases of CIN during recent years. For many years, gadolinium-based contrast agents have been considered as safe, but in 2006 the first reporting of patients who had developed a new rare potentially fatal disease called NSF in the weeks after exposure to gadolinium-based contrast agents began. However, it was not until 2006 that the NSF was linked to gadolinium contrast agents and it was proposed that the free gadolinium from the contrast agent could be a trigger for NSF. NSF is a connective tissue disease which usually manifests itself as a skin disease with swelling in arms and legs, but can also affect internal organs. NSF occurs in combination with chronic kidney disease and has only recently been particularly investigated.

Therefore, it is essential to clarify if these reactions are actually directly related to the application of contrast agents or to MR/CT-examinations. Most major studies conducted on gadolinium-based and iodine-containing contrast agents have been retrospective, and so far no similar large scale study has been performed independently from pharmaceutical companies. Thus, there is a lack of independent studies, which investigate the severity of adverse reactions as well as delayed adverse reactions one month after the patients have been exposed to the contrast agent.The study aim is to investigate the safety profile for respectively iodine-containing and gadolinium-based contrast agents to CT and MR- examinations in a prospective design. A control group examined without the use of contrast agent will be included, so that the study can illuminate reported adverse reactions related to contrast agents and CT/MR-examinations. This applies to renal, non-renal, and late adverse reactions.

This project will ultimately illuminate any significant and life-threatening late effects and therefore, these will be detected earlier, and it will become more likely to treat the patients in good time for these events. The following series of hypotheses will be investigated in this study:

1. Renal as well as non-renal adverse reactions occurring are related to the use of contrast agent in MR-/CT-examination.
2. CIN occurs in patients undergoing a MR-/CT-examination with contrast agent.

Methods:

Approvals from The Copenhagen County Committee on Biomedical Research Ethics and The Danish Data Protection Agency are obtained. The study will be conducted as a prospective study at Herlev Hospital, Department of Radiology. Patients referred to an MR/CT-examination will be offered participation in the study. Since the patients are referred to a MR-/CT-examination as part of their patient diagnostic evaluation, the distribution into different groups will be without any influence from the study officials.The study includes a total of 1600 patients in a period of approximately 2 years. The patients will be distributed in four groups (a, b, c and d) with 400 patients in each group. Group a and c (case group) undergo respectively MR- and CT- examinations with respectively gadolinium-based contrast agent and iodine-containing contrast agent. Group b and d (control groups) will undergo MR/CT-examination without any use of contrast agent. Informed consent will be obtained from all patients. Data will be collected continuously. For each participating patient the following will be registered: risk factors (patients allergic to gadolinium-based and iodine-containing contrast agents, patients with renal impairment and diabetes), estimated kidney function (eGFR) with a finger stick blood test immediately before and 72 hours after the MR/CT-examination. The blood test is quick, easy and requires no more than a small stick on the side of the finger tip with a finger stick. The blood drop is placed on a test strip and into a renal function meter, whereupon eGFR is read. The test strip will be destroyed immediately after completion of the test/ measurement. To detect the occurrence of acute adverse reactions after administration of contrast agents, the patients are observed for 30 min. Patients in the control groups will also be observed for 30 minutes after start of MR/CT-examination. All patients are supplied with two questionnaires regarding the occurrence of adverse reactions and possible delayed reactions, which they must complete 72 hours and one month after MR/CT-examination. Results from group a will be compared with results from group b, while the results from group c will be compared with results from group d. This study will not be statistically randomized, since it is an observational study. Furthermore, it is necessary to have a major control group.

Adverse reactions, risks and disadvantages:There are no known adverse reactions in this study, when the exclusion criteria are met. Patients will already be referred for an MR/CT- examination, and contrast agents that are already approved by health authorities will be used as tools for MR/CT-examinations. Therefore, this study does not pose a greater risk or inconvenience to the participants. Moreover, there are no adverse reactions associated with the blood tests measurement.

Economic conditions:

Study officials have no financial ties to private firms or pharmaceutical companies with interest in this study. Since the majority of researches on contrast agents are made by pharmaceutical companies, this project is important and of great interest since it is independent from the pharmaceutical industry. Therefore, the project's conclusions will not be influenced by strategic and economic interests.

Ethical considerations:

This study is unique in the sense that it so far is, the only major prospective study that follows patients one month after completion of MR/CT-examination. The study is primarily intended as a method to clarify the extent of late adverse reactions that may occur after the patient has left the examination room. For precisely these contrast agents, it is advantageous to have a study which provides a comprehensive systematic overview of acute and late adverse reactions, because many severe and life-threatening late adverse reactions occur days and even weeks after the contrast agent administration. We hope that this study will result in an improved documentation of whether the incidences of acute and delayed severe adverse reactions are directly related to the use of contrast agents for MR/CT-examinations. This will increase patient safety because; it will help clarifying whether adverse reactions are related to contrast agents or MR/CT-examination. For the individual participant the benefit of participation in this study means that, in future any significant delayed adverse reaction will be discovered in time. Furthermore, a detection of the presence of mild or/and moderate adverse reactions will lead to, an earlier treatment of these adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred to a MR/CT-examination at Herlev Hospital, Department of Radiology
* Age > 18 years

Exclusion Criteria:

* Age < 18 years
* Increased metabolism (hyperthyroidism)
* Dementia
* Pregnancy / lactation
* Patients who have undergone MR/CT- examinations within the last month prior to the actual examination
* New MR/CT-examination (enhanced and unenhanced) in the observation period (one month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from Herlev Hospital, Department of Radiology. Patients referred to an MR/CT-examination will be offered participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1467 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Renal and non-renal adverse events to enhanced and unenhanced CT and MRI | before, 3 days and 1 month after enhanced or unenhanced CT and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Manal Azzouz, MSc Pharmacy, Principal Investigator — Department of Diagnostic Radiology,Copenhagen University Hospital Herlev; Henrik S Thomsen, Study Director — Department of Diagnostic Radiology,Copenhagen University Hospital Herlev
Locations (1):
- Department of Diagnostic Radiology,Copenhagen University Hospital Herlev, Herlev, Denmark

REFERENCES:
- [Background] Weinreb JC. Which study when? Is gadolinium-enhanced MR imaging safer than iodine-enhanced CT? Radiology. 2008 Oct;249(1):3-8. doi: 10.1148/radiol.2493200803. No abstract available. PMID 18796663
- [Background] Hunt CH, Hartman RP, Hesley GK. Frequency and severity of adverse effects of iodinated and gadolinium contrast materials: retrospective review of 456,930 doses. AJR Am J Roentgenol. 2009 Oct;193(4):1124-7. doi: 10.2214/AJR.09.2520. PMID 19770337
- [Background] Morcos SK. Review article: Acute serious and fatal reactions to contrast media: our current understanding. Br J Radiol. 2005 Aug;78(932):686-93. doi: 10.1259/bjr/26301414. PMID 16046418
- [Background] Remy-Jardin M, Dequiedt P, Ertzbischoff O, Tillie-Leblond I, Bruzzi J, Duhamel A, Remy J. Safety and effectiveness of gadolinium-enhanced multi-detector row spiral CT angiography of the chest: preliminary results in 37 patients with contraindications to iodinated contrast agents. Radiology. 2005 Jun;235(3):819-26. doi: 10.1148/radiol.2353040734. Epub 2005 Apr 21. PMID 15845797
- [Background] Cutroneo P, Polimeni G, Curcuruto R, Calapai G, Caputi AP. Adverse reactions to contrast media: an analysis from spontaneous reporting data. Pharmacol Res. 2007 Jul;56(1):35-41. doi: 10.1016/j.phrs.2007.03.003. Epub 2007 Mar 25. PMID 17482832
- [Background] Hosoya T, Yamaguchi K, Akutsu T, Mitsuhashi Y, Kondo S, Sugai Y, Adachi M. Delayed adverse reactions to iodinated contrast media and their risk factors. Radiat Med. 2000 Jan-Feb;18(1):39-45. PMID 10852654
- [Background] Ledneva E, Karie S, Launay-Vacher V, Janus N, Deray G. Renal safety of gadolinium-based contrast media in patients with chronic renal insufficiency. Radiology. 2009 Mar;250(3):618-28. doi: 10.1148/radiol.2503080253. PMID 19244037
- [Background] Dillman JR, Ellis JH, Cohan RH, Strouse PJ, Jan SC. Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol. 2007 Dec;189(6):1533-8. doi: 10.2214/AJR.07.2554. PMID 18029897
- [Background] Grobner T. Gadolinium--a specific trigger for the development of nephrogenic fibrosing dermopathy and nephrogenic systemic fibrosis? Nephrol Dial Transplant. 2006 Apr;21(4):1104-8. doi: 10.1093/ndt/gfk062. Epub 2006 Jan 23. No abstract available. PMID 16431890
- [Background] Marckmann P, Skov L, Rossen K, Dupont A, Damholt MB, Heaf JG, Thomsen HS. Nephrogenic systemic fibrosis: suspected causative role of gadodiamide used for contrast-enhanced magnetic resonance imaging. J Am Soc Nephrol. 2006 Sep;17(9):2359-62. doi: 10.1681/ASN.2006060601. Epub 2006 Aug 2. PMID 16885403
- [Background] Schild HH, Kuhl CK, Hubner-Steiner U, Bohm I, Speck U. Adverse events after unenhanced and monomeric and dimeric contrast-enhanced CT: a prospective randomized controlled trial. Radiology. 2006 Jul;240(1):56-64. doi: 10.1148/radiol.2393050560. Epub 2006 May 23. PMID 16720865
- [Derived] Azzouz M, Romsing J, Thomsen HS. Fluctuations in eGFR in relation to unenhanced and enhanced MRI and CT outpatients. Eur J Radiol. 2014 Jun;83(6):886-892. doi: 10.1016/j.ejrad.2014.02.014. Epub 2014 Feb 24. PMID 24656402
- [Derived] Azzouz M, Romsing J, Thomsen HS. Can a structured questionnaire identify patients with reduced renal function? Eur Radiol. 2014 Mar;24(3):780-4. doi: 10.1007/s00330-013-3065-x. Epub 2013 Nov 26. PMID 24275804